CLINICAL TRIAL: NCT05445869
Title: A Prospective, Multi-Center, Single-Arm, Open-Label, Observational Study on the Safety and Effectiveness of the ProSomnus EVO Sleep and Snore Device in the Treatment of Severe Obstructive Sleep Apnea
Brief Title: Severe OSA Study (SOS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated by Sponsor.
Sponsor: ProSomnus Sleep Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PST202101
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Obstructive Sleep Apnea; Sleep Apnea
Keywords: oral appliance; mandibular advancement device
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- EVO Sleep and Snore Device (Experimental): Participants will be provided with a custom EVO Sleep and Snore Device
  Interventions: Device: ProSomnus® EVO Sleep and Snore Device

INTERVENTIONS:
Device: ProSomnus® EVO Sleep and Snore Device — The ProSomnus® EVO Sleep and Snore Device is an intraoral device for snoring and obstructive sleep apnea. It works by repositioning the mandible during sleep, thereby improving the flow of air through the patient's pharyngeal space. The ProSomnus® EVO Sleep consists of maxillary and mandibular device arches that are CAD/CAM designed with twin-mated posts and digitally milled to be patient-specific according to physician prescription. Prescribed advancements can be achieved by simply removing the current upper or lower device arch and inserting the next upper or lower device arch in the mandibular advancement series. The device does not have any adjustment mechanisms to modify or maintain the mandibular position such as pistons, screws, straps, or repositioning elastics. The device is supplied nonsterile.

SUMMARY:
This study is a prospective, multi-center, single-arm, open-label study evaluating the safety and effectiveness of therapy with the ProSomnus EVO Sleep and Snore Device in individuals with severe obstructive sleep apnea.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, single-arm, open-label study evaluating the safety and effectiveness of therapy with the ProSomnus EVO Sleep and Snore Device in individuals with severe obstructive sleep apnea (OSA). Study participants will receive a custom ProSomnus EVO Sleep and Snore device and then be tested using a Type II home sleep apnea test (HSAT) to determine if they have achieved apnea-hypopnea index (AHI) < 15 h-1 with the device in place. Home sleep apnea testing will be conducted at predetermined timepoints rather than based on subjective measures such as symptom alleviation. After completing a set device advancement and testing protocol, study participants will complete a final HSAT six months after therapy initiation. This value will be used to determine the therapeutic success rate of the appliance. Safety evaluations will be conducted at each study visit that takes place after therapy initiation. These evaluations, along with dental examinations and adverse event reports, will be used to determine if the safety endpoint is met. Participants will continue to be followed for an additional six months after collection of data for the primary endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, of any race, aged 18-80 years (inclusive)
4. Diagnosed with uncomplicated severe OSA (i.e., AHI > 30 h-1); where uncomplicated is defined by the absence of:

   1. Conditions that place the patient at increased risk of non-obstructive sleep-disordered breathing (e.g., central sleep apnea, hypoventilation, and sleep-related hypoxemia). Examples of such conditions include significant cardiopulmonary disease, potential respiratory muscles weakness due to neuromuscular conditions, history of stroke, and chronic opiate medication use.
   2. Concern for significant non-respiratory sleep disorder(s) that require evaluation (e.g., disorders of central hypersomnolence, parasomnias, sleep-related movement disorders) or interfere with accuracy of HSAT (e.g., severe insomnia).
   3. Environmental or personal factors that preclude the adequate acquisition and interpretation of data from HSAT.
5. Body mass index (BMI) < 40 kg/m2
6. Neck circumference < 50 cm
7. Absence of severe oxyhemoglobin desaturation during sleep, indicated by mean nocturnal SpO2 > 87%
8. Mandibular range of motion > 5 mm in protrusive direction
9. Adequate dentition, as determined by the site dentist

Exclusion Criteria:

1. Inability to breathe through the nose comfortably
2. Presence of > 25% CSA
3. Presence of positional obstructive sleep apnea per Cartwright's definition32
4. History of surgery intended to alter anatomy for the correction of OSA, such as uvulopalatopharyngoplasty (UPPP), maxillomandibular advancement (MMA), or tongue/hyoid suspension. History of surgery intended to restore normal anatomy, such as tonsillectomy, adenoidectomy, septoplasty, or polypectomy, is permitted
5. Presence of hypoglossal nerve stimulation device
6. Use of CPAP or OAT within the two weeks prior to the screening HSAT
7. History of OAT that has been demonstrated to provide effective therapy within the two years prior to the screening HSAT
8. Anticipated change in medical therapy during the study protocol that could alter OSA severity (e.g., weight loss surgeries; UPPP, MMA, tongue/hyoid suspension)
9. Loose teeth or advanced periodontal disease
10. History of temporomandibular joint disorder
11. Resistant hypertension, defined as inadequately controlled blood pressure despite therapy with ≥ 3 oral hypertensive agents
12. Presence of congestive heart failure, recurrent atrial fibrillation, or coronary artery disease
13. Presence of neuromuscular diseases, hypoventilation disorders, or cerebrovascular disease
14. Presence of pulmonary disease resulting in significant desaturation, e.g., severe chronic obstructive pulmonary disease, interstitial lung disease (SaO2 nadir of 87%), or pulmonary hypertension
15. History of cerebrovascular incident within the last 12 months
16. Use of pacemaker or other life supporting device
17. Anticipated change in body weight > 5% during the study period
18. Participation in other studies that could interfere with the study protocol
19. Pregnancy or lactation
20. In the opinion of the investigator, unsuitable for inclusion in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Efficacy (apnea-hypopnea index) | 6 months
  The AHI co-primary effectiveness endpoint is to demonstrate a responder rate significantly greater than 50%; responders will be defined as individuals who achieve an AHI < 15 h-1 with the EVO Sleep and Snore Device 6 months after initiation of the therapy.
Efficacy (oxygen desaturation index) | 6 months
  The ODI co-primary effectiveness endpoint is to demonstrate a responder rate significantly greater than 50%; responders will be defined as individuals who achieve decrease in ODI from baseline of 25% or more with the EVO Sleep and Snore Device 6 months after initiation of the therapy.
Evaluation of safety (adverse events, dental examinations, safety examinations) | 6 months
  The primary safety endpoint is to demonstrate an acceptable safety profile of the EVO Sleep and Snore Device, determined through assessment of all reported adverse events, dental examinations, and safety evaluations. There will be no formal statistical analysis.

SECONDARY OUTCOMES:
Epworth Sleepiness Scale | 6 months
  The secondary endpoint is to demonstrate that the minimum clinically important difference (MCID) of -2 on the Epworth Sleepiness Scale (ESS) is achieved in participants with moderate to excessive daytime sleepiness (defined as ESS > 12). The Epworth Sleepiness Scale is a scale that ranges from 0 (no daytime sleepiness) to 18 (excessive daytime sleepiness).

CONTACTS AND LOCATIONS:
Overall Officials: Erin Mosca, PhD, Study Director — ProSomnus Sleep Technologies
Locations (5):
- United States (5):
  - Stanford Sleep Medicine Clinic, Redwood City, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Advanced ENT Physicians and Surgeons of CNY, Fayetteville, New York
  - Mount Sinai Integrative Sleep Center, New York, New York